CLINICAL TRIAL: NCT05628246
Title: Telemedicine Improves Pain-related Disabilities in Following up Cancer Pain Outpatient: A Prospective Non-randomized Study.
Brief Title: Telemedicine Improves Pain-related Disabilities in Following up Cancer Pain Outpatient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Si 310/2022
Record Dates: First submitted 2022-11-15; First posted 2022-11-28 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Pain, Chronic; Cancer Pain
MeSH Terms: conditions — Chronic Pain; Cancer Pain | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person (Active Comparator): Face to face at OPD
  Interventions: Other: In-person
- Telemedicine (Experimental): Telemedicine
  Interventions: Other: Telemedicine

INTERVENTIONS:
Other: Telemedicine — Telemedicine
  Arms: Telemedicine
Other: In-person — In-person
  Arms: In-person

SUMMARY:
Cancer is the second leading cause of death worldwide, with approximately 18.1 million new cases and 9.6 million deaths reported in 2018. Cancer-related pain is experienced by 50-70% of patients, with a higher prevalence at advanced disease stages (66.4%). Since the development of WHO's cancer pain guidelines, several studies have reported good relief of symptoms and suffering for a majority of patients. Recent reports suggest that up to 50% of patients still report insufficient pain control. Patients with cancer often present with multiple symptoms and functional decline. Evidence supports multidisciplinary approaches to address symptoms and suffering, including early palliative care referral

From review literatures we found that the telemedicine group had significantly higher quality of life than the usual care group. In addition, the telemedicine group had lower anxiety and depression scores than the usual care group.

Therefore, we will conduct the non-randomized controlled study of using telemedicine comparing to conventional in-person at OPD in hospitalized cancer pain patients.

The purpose of this study is to assess the pain interference by using the Brief Pain Inventory (BPI) and to compare between the in-person group and the telemedicine group. To assess the cost-effectiveness of telemedicine for reducing symptoms associated with cancer and its treatment.

DETAILED DESCRIPTION:
The pain interference will be assessed and compared using Brief Pain Inventory from 0-70 between In-person group and telemedicine group at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years old
* Cancer patients who new visit as out patient at pain clinic, Siriraj hospital

Exclusion Criteria:

* Cannot read and write
* Confusion
* Unable to use the 0-10 Numerical Rating Scale (NRS) to rate pain intensity.
* Unstable clinical presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2025-07-17 (Estimated); Study Completion 2025-07-17 (Estimated)

PRIMARY OUTCOMES:
Pain interference | at 1 month
  The pain interference will be assessed and compared using Brief Pain Inventory from 0-70 between In-person group and telemedicine group.

SECONDARY OUTCOMES:
Quality of life (QoL) | at 1 month
  The quality of life will be assessed and compared using EuroQoL 5D5L between In-person group and telemedicine group.
Pain intensity | at 1 month, 2 months and 3 months
  The pain reduction will be assessed and compared using numerical rating (NRS) from 0-10; 0 designating "no pain" and 10 designating " worst possible pain" scale between In-person group and telemedicine group.

CONTACTS AND LOCATIONS:
Overall Officials: Suratsawadee Wangnamthip, M.D., Study Director — Mahidol University
Locations (1):
- Faculty of medicine Siriraj Hospital Mahidol University, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pang L, Liu Z, Lin S, Liu Z, Liu H, Mai Z, Liu Z, Chen C, Zhao Q. The effects of telemedicine on the quality of life of patients with lung cancer: a systematic review and meta-analysis. Ther Adv Chronic Dis. 2020 Oct 7;11:2040622320961597. doi: 10.1177/2040622320961597. eCollection 2020. PMID 33101621
- [Result] Wangnamthip S, Panchoowong S, Donado C, Lobo K, Phankhongsap P, Sriveerachai P, Euasobhon P, Rushatamukayanunt P, Mandee S, Zinboonyahgoon N, Berde CB. The Effectiveness of Cancer Pain Management in a Tertiary Hospital Outpatient Pain Clinic in Thailand: A Prospective Observational Study. Pain Res Manag. 2021 Jul 20;2021:5599023. doi: 10.1155/2021/5599023. eCollection 2021. PMID 34336068
- [Result] Chaudakshetrin P. Validation of the Thai Version of Brief Pain Inventory (BPI-T) in cancer patients. J Med Assoc Thai. 2009 Jan;92(1):34-40. PMID 19260241
- [Result] Pattanaphesaj J, Thavorncharoensap M, Ramos-Goni JM, Tongsiri S, Ingsrisawang L, Teerawattananon Y. The EQ-5D-5L Valuation study in Thailand. Expert Rev Pharmacoecon Outcomes Res. 2018 Oct;18(5):551-558. doi: 10.1080/14737167.2018.1494574. Epub 2018 Jul 6. PMID 29958008